## STATISTICAL ANALYSIS PLAN

Study Title: Early Community Client-Led ART Delivery (CCLAD) to Optimize HIV Care Engagement in Nakivale Refugee Settlement

Document Date: 31 March 2023

NCT04736316

## STATISTICAL ANALYSIS PLAN

Counts and frequencies were reported for demographic characteristics, mental health conditions (depression, anxiety, PTSD), self-reported health status, and social support for the overall sample and were stratified by Early CCLAD participation. Among Early CCLAD participants, the proportions of those who initiated ART, and the proportion who became virally suppressed were documented. Additionally, among Early CCLAD participants, the number of visits with Early CCLAD groups and HIV clinic visits were recorded.